CLINICAL TRIAL: NCT07061821
Title: Evaluation of Left Ventricular Ejection Fraction Using an Accelerated Cardiac Cine-MRI Sequence With Deep Learning-based Image Reconstructions Compared to the Reference Cine-MRI Sequence in the Assessment or Follow-up of Left Ventricular Hypertrophy
Brief Title: Evaluation of Left Ventricular Ejection Fraction Using an Accelerated Cardiac Cine-MRI Sequence With Deep Learning-based Image Reconstructions
Acronym: HVGLD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2025_843_0122
Record Dates: First submitted 2025-07-01; First posted 2025-07-11 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Left Ventricular Ejection Fraction; Cardiac Magnetic Resonance Imaging; Deep Learning; Image Reconstruction; Left Ventricular Hypertrophy
Keywords: Left Ventricular Hypertrophy; Left Ventricular Ejection Fraction; Cardiac Magnetic Resonance Imaging; Deep Learning; Image Reconstruction
MeSH Terms: conditions — Hypertrophy, Left Ventricular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: accelerated cardiac cine-MRI sequence — Addition of an accelerated cardiac cine-MRI sequence with deep learning-based image reconstruction to the standard cardiac MRI protocol, performed during the same session

SUMMARY:
Left ventricular hypertrophy (LVH) is a common condition that may result from hypertension, hypertrophic cardiomyopathy, aortic valve stenosis, or certain metabolic disorders. Cardiac imaging is essential for diagnosis, prognostic assessment, and quantification of cardiac function. While transthoracic echocardiography remains widely used, it is limited by acoustic window dependence and inter-observer variability. Cardiovascular Magnetic Resonance (CMR) imaging currently serves as the reference standard for measuring left ventricular ejection fraction (LVEF), cardiac volumes, and tissue characterization. However, conventional cine-CMR sequences require repeated breath-holds, which are often challenging for elderly or dyspneic patients, generating respiratory motion artifacts that compromise image quality. Accelerated cine-CMR sequences with deep learning-based image reconstructions offer a promising alternative by significantly reducing acquisition time while preserving image quality. This study aims to evaluate whether these accelerated cine-CMR sequences provide LVEF measurements concordant with conventional cine-CMR sequences, with potential to improve patient comfort and reduce examination time.

ELIGIBILITY:
Inclusion Criteria:

* Patient referred for cardiac MRI as part of the assessment or follow-up of left ventricular hypertrophy
* Age ≥ 18 years old
* Ability of the subject to understand and express his consent
* Affiliation to the social security scheme

Exclusion Criteria:

* Severe obesity (>140 kg) preventing the patient from entering the scanner bore, which has a diameter of less than 70 cm
* Age ≥ 18 years old
* Person under guardianship or curators, or deprived of liberty
* Pregnant or breastfeeding woman
* Known allergy to gadolinium chelates
* Claustrophobia
* Any contraindication to MRI
* Arrhythmia
* Inability to hold breath for more than 10 seconds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
LVEF Difference between both sequences | day 1
  Value of the difference between the measurement of left ventricular ejection fraction (LVEF) obtained using the accelerated cardiac cine-MRI sequence with Deep Learning-based image reconstruction compared to the conventional cine-MRI sequence.

SECONDARY OUTCOMES:
difference of end-diastolic volume of the left ventricle between both sequences | day 1
  Value of the difference between the measurements of end-diastolic volumes of the left ventricle obtained using the accelerated cardiac cine-MRI sequence with Deep Learning-based image reconstruction compared to the conventional cine-MRI sequence.
difference of end-systolic volume of the left ventricle between both sequences | day 1
  Value of the difference between the measurements of end-systolic volumes of the left ventricle obtained using the accelerated cardiac cine-MRI sequence with Deep Learning-based image reconstruction compared to the conventional cine-MRI sequence.
Differnce of measurement of the global longitudinal strain of the left ventricle between both sequences | day 1
  Value of the difference between the measurement of global longitudinal strain of the left ventricle obtained using the accelerated cardiac cine-MRI sequence with Deep Learning-based image reconstruction compared to the conventional cine-MRI sequence.
Difference of the left ventricular mass between both sequences | day 1
  Value of the difference between the measurement of left ventricular mass obtained using the accelerated cardiac cine-MRI sequence with Deep Learning-based image reconstruction compared to the conventional cine-MRI sequence.
diffrence of the maximal thickness of the left ventricle between both sequences | day 1
  Value of the difference between the measurement of maximal thickness of the left ventricle obtained using the accelerated cardiac cine-MRI sequence with Deep Learning-based image reconstruction compared to the conventional cine-MRI sequence.
Difference of the acquisition time between both sequences | day 1
  Value of the difference in acquisition time between the accelerated cardiac cine-MRI sequence with Deep Learning-based image reconstruction and the conventional cine-MRI sequence

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No